CLINICAL TRIAL: NCT06428994
Title: Risk for Subsequent Osteoradionecrosis in A Transferred Fibula Flap in Head and Neck Cancer Patients Undergoing Segmental Mandibulectomy: a Cohort Study
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: No. 201800172B0
Record Dates: First submitted 2024-05-12; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2018-02

CONDITIONS: Head and Neck Cancer; Fibula Flap; Osteoradionecrosis; Mandibulectomy
MeSH Terms: conditions — Head and Neck Neoplasms; Osteoradionecrosis | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ORN: ORN in this study is defined as exposed irradiated bone tissue that fails to heal over a period of three months without residual or recurrent tumors.
  Interventions: Radiation: Radiotherapy
- non-ORN: Patients without ORN.

INTERVENTIONS:
Radiation: Radiotherapy — Post-operative radiotherapy for head and neck cancer
  Groups: ORN

SUMMARY:
A retrospective analysis of 329 patients at one single institution between January 2014 and December 2019 who underwent free fibula flap reconstruction was conducted. A variety of clinicopathological postoperative parameters were identified and assessed.

DETAILED DESCRIPTION:
The study was conducted as a monocentric, retrospective study. Patients who underwent a mandibular reconstruction with a free fibula flap due to head and neck cancer through January 2014 to December 2019 at one single institution in Taiwan were identified. All charts including surgical records, progress notes, nursing records, clinic notes, imaging study after surgery were reviewed. Data extraction was performed for the following variables: Patient demographics, primary diagnosis, cancer location and staging, treatment prior to index surgery, postoperative hemoglobin and albumin, operating time, flap type, mandibular defect length, type of the defect according to Jewer's classification, ischemia time, number of fibula segments, plate type, re-exploration, time of hospitalization, postoperative radiotherapy and/or chemotherapy, ORN cases, identification time of ORN and management for ORN. The patients were then organized into two groups: ORN and non-ORN. This research was approved by the Institutional Review Board of our hospital (No. 201800172B0), which was available until 2022/02/28. The investigators completed data analysis before 2022/02/28 and then initiated manuscript preparing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a mandibular reconstruction with a free fibula flap due to head and neck cancer through January 2014 to December 2019.

Exclusion Criteria:

* Cases with incomplete medical records.
* Patients who did not attend at least 6 months of follow ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2014 and December 2019, 580 patients received free fibula flap mandibular reconstruction, with 374 of them attributed to head and neck cancer reconstruction. Cases with incomplete medical records were excluded (n = 9). Additionally, patients who did not attend at least 6 months of follow-up were also excluded (n = 36). Finally, 329 patients including 309 males and 20 females met the inclusion criteria of this study.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence on development osteoradionecrosis(ORN) in free fibula flaps | Up to 7 years postoperatively
  The incidence of osteoradionecrosis in patients who received free fibula flap reconstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Angela Chien-Yu Chen, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No